CLINICAL TRIAL: NCT06744010
Title: Sub Sartorial Canal Block and Popliteal Block Versus Femoral Block and Popliteal Block in Ankle Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Safaa Gaber Ragab, Associate professor of anaethesiology, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: M 739
Record Dates: First submitted 2024-12-12; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Sub Sartorial Canal Block and Popliteal Block Versus Femoral Block and Popliteal Block in Ankle Surgeries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): sub sartorial canal block + popliteal block
  Interventions: Procedure: Sub sartorial canal block and popliteal block in ankle surgeries
- Group B (Experimental): femoral block + popliteal block
  Interventions: Procedure: femoral block and popliteal block in ankle surgeries

INTERVENTIONS:
Procedure: Sub sartorial canal block and popliteal block in ankle surgeries — All patients will be anesthetized with PNBs for surgery.
  * PNBs will be performed in a block room at least 30minute preoperatively.
  * All PNBs will be performed under ultrasound guidance (LOGIQ P6, GE Healthcare; Chicago, IL) using a high-frequency linear transducer (3.4-10.8MHz).
  * All blocks will be performed after skin preparation with 2% chlorhexidine gluconate by 1 orthopedic surgeon (YUP) with vast experience in ultrasound-guided nerve block techniques.
  * A 22-ga Tuohy needle will be introduced in-plane and 2 to 3mL of saline will be used to confirm the correct position of the needle tip near the target nerve.
  * The study medication will be administered through the needle as a bolus of 20mL of a 1:1 mixed solution of bupivacaine 0.75% and lidocaine 1%.
  * The total volume per every block will be 20 ml in the form of bupivacaine 1.25% with 1:200,000 epinephrine and 250 mg Mgso4.
  Arms: Group A
Procedure: femoral block and popliteal block in ankle surgeries — * All patients will be anesthetized with PNBs for surgery.
  * PNBs will be performed in a block room at least 30minute preoperatively.
  * All PNBs will be performed under ultrasound guidance (LOGIQ P6, GE Healthcare; Chicago, IL) using a high-frequency linear transducer (3.4-10.8MHz).
  * All blocks will be performed after skin preparation with 2% chlorhexidine gluconate by 1 orthopedic surgeon (YUP) with vast experience in ultrasound-guided nerve block techniques.
  * A 22-ga Tuohy needle will be introduced in-plane and 2 to 3mL of saline will be used to confirm the correct position of the needle tip near the target nerve.
  * The study medication will be administered through the needle as a bolus of 20mL of a 1:1 mixed solution of bupivacaine 0.75% and lidocaine 1%.
  * The total volume per every block will be 20 ml in the form of bupivacaine 1.25% with 1:200,000 epinephrine and 250 mg Mgso4.
  Arms: Group B

SUMMARY:
Ankle surgeries are severely painful. A sciatic nerve block is typically not enough to cover the pain sources (Delbos et al., 2019).

It can be speculated that approaching the saphenous nerve in the subsartorial compartment distal to the point where it pierces the vastoadductor membrane but proximal to the point where it penetrates the crural fascia and becomes subcutaneous would selectively target the saphenous nerve without any decrease of quadriceps strength (Jensen et al., 2024).

Previous study showed that femoral nerve block (FNB) provides good surgical anesthesia and good postoperative pain control for patients with ankle conditions (Lee et al., 2014). However, FNB leads to femoral quadriceps muscle weakness (Jaeger et al., 2013).

Consequently, quadriceps weakness results in functional impairment and it is associated with an increased risk of postoperative falls (Johnson et al., 2013).

Thus far, attempts to reduce quadriceps involvement after FNB without compromising analgesia have not been successful (Li et al., 2019).

Partially because of the increase in the use of ultrasound guidance, a more targeted approach that only blocks sensory fibers of the femoral nerve that supply the operative site has been attempted; thus, the feasibility of sub sartorial canal block has been studied (Kopp et al., 2017).

In recent years, sub sartorial canal block has been successfully used for postoperative pain control after knee surgery (Lavand'homme et al., 2022).

However, no randomized, control study has compared sub sartorial canal block to femoral nerve block for ankle surgeries. We hypothesized that compared to femoral nerve block, sub sartorial canal block would demonstrate noninferior pain scores during surgery and until 48 hours postoperatively and cause less weakness in the quadriceps.

DETAILED DESCRIPTION:
Sample size was calculated using Power Analysis and Sample Size Software (PASS 2020) "NCSS, LLC. Kaysville, Utah, USA, ncss.com/software/pass". Based on a previously published study (Lavand'homme et al., 2022) and (Joe et al., 2016); the VAS pain scores of the adductor canal block group were not inferior during and after the operation compared to those of the FNB group. At 30 minutes and 2 hours after anesthesia, patients who received an adductor canal block had significantly higher average dynamometer readings than those who received a FNB (34.2±20.4 and 30.4±23.7 vs 1.7±3.7 and 2.3±7.4, respectively), and the results were similar at 24 and 48 hours after anesthesia. Based on this, a minimal total hypothesized sample size of 60 eligible patients will be needed taking into consideration 95% level of confidence, an effect size of 1/100 and 5% margin of error using two-sided proportional Z- test. Sample size will be increased 20% for possible dropout rate, so 72 patients will be enrolled in the study (36 in each group).

* Randomization: It will be based on a computer-generated block randomization list (4 numbers per block) in a 1:1 ratio. All patients underwent sub sartorial canal block + popliteal block, or femoral block + popliteal block according to a randomized assignment . the randomization sequence was kept hidden in sealed opaque envelopes. After recruitment and admittance to blocking room , the authors unwrapped the envelopes . the allocations of the group were blinded to assessors , data collectors with an expert anesthesiologist doing the block (single blinded).
* Study tools:

  1. After approval of study protocol, patients will be enrolled into the study according to inclusion and exclusion criteria.
  2. A total of 72 patients will be categorized into 2 groups:

     * Group A "sub sartorial canal block + popliteal block".
     * Group B "femoral block + popliteal block".
  3. Anesthesia and postoperative analgesia:

     * All patients will be anesthetized with PNBs for surgery.
     * PNBs will be performed in a block room at least 30minute preoperatively.
     * All PNBs will be performed under ultrasound guidance (LOGIQ P6, GE Healthcare; Chicago, IL) using a high-frequency linear transducer (3.4-10.8MHz).
     * All blocks will be performed after skin preparation with 2% chlorhexidine gluconate by 1 orthopedic surgeon (YUP) with vast experience in ultrasound-guided nerve block techniques.
     * A 22-ga Tuohy needle will be introduced in-plane and 2 to 3mL of saline will be used to confirm the correct position of the needle tip near the target nerve.
     * The study medication will be administered through the needle as a bolus of 20mL of a 1:1 mixed solution of bupivacaine 0.75% and lidocaine 1%.
     * The total volume per every block will be 20 ml in the form of bupivacaine 1.25% with 1:200,000 epinephrine and 250 mg Mgso4.
     * For the ultrasound-guided sub sartorial compartment block of the saphenous nerve, the patient will be placed in the supine position with external rotation of the thigh and slight flexion of the knee. A 15 MHz linear ultrasound probe (PX, FUJIFILM SonoSite, Bothell, Washington, USA) will be placed in the transverse plane across the sartorius muscle approximately at the base of the patella. The sartorius muscle will be followed proximally and distally in order to visualize the segment of the sub sartorial compartment between the two points where the saphenous nerve intersected the tendons of the adductor magnus and semimembranosus muscles, respectively. The saphenous nerve will be visualized in the proximal half of this segment of the subsartorial compartment - just distal to the intersection of the saphenous nerve and the tendon of the adductor magnus muscle. At this level there is a well-defined subsartorial compartment between the sartorius muscle tendon and the so-called 'subsartorial fat pad' that is compliant for injection. The needle will be inserted ultrasound-guided in-plane from anterior to posterior and advanced in order to place the needle tip adjacent to the saphenous nerve and inject perineurally.
     * For popliteal sciatic nerve block, the patient will be lain laterally on the opposite side of the limb which has to be blocked. The limb to be blocked will be flexed partially at hip and knee joint. Using a high-frequency linear probe, a scan of popliteal fossa will be conducted to identify separate tibial and common peroneal nerves lying superficially and posteriorly to popliteal artery. Movement of the probe proximally brings tibial and common peroneal nerves together to form the sciatic nerve at a variable point, above the popliteal crease. At this level, via out-of plane technique, using 21 gauge insulated needle, 20 ml of 0.5% ropivacaine will be deposited after negative aspiration and real-time spread of local anesthetic will be visualized in sub paraneural space around the sciatic nerve.
     * For the femoral nerve block, the femoral nerve will be identified lateral to the femoral artery at the inguinal crease in the transverse section. The study medication will be injected anterior and posterior to the nerve.
  4. The actual or estimated needle insertion sites will be covered with a dressing bandage in all patients to blind those assessing the outcome of the procedure to the treatment.
  5. Intravenous ketorolac tromethamine (30mg, maximum dose 90mg/d) will be given as a rescue analgesic during the first 48 hours postoperatively when a patient reported a visual analog scale (VAS) score of ≥5 or if the patient requested pain relief.
  6. All the patients will receive 0.03 mg/kg of intra-venous midazolam and oxygen will be supplied by face mask throughout the procedure.
  7. Surgery will be started after adequate sensory and motor blockade will be achieved.
  8. In patients with failure to achieve adequate surgical anesthesia after 20 minutes of administration of block, it will be considered as a block failure and converted to general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult patients who will be scheduled to undergo surgery on medial side of the ankle, or both sides of the ankle (Achilles tendon surgery, the removal of an implanted device on the medial side, or ankle arthroscopy) under peripheral nerve blocks (PNBs).

  2. Patients have an American Society of Anesthesiologists Physical status of I to II.

  3. Age 19 to 65 years.

Exclusion Criteria:

- 1. An inability of patient to cooperate. 2. A history of alcohol or drug abuse. 3. Those with rheumatoid arthritis, coagulation disorders, peripheral neuropathy.

4. Known allergies to local anesthetics. 5. Recent use of opioids, corticosteroids, or any other analgesics. 6. If a patient complained of incomplete block before the end of surgery, we will exclude the patient from the analysis.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Visual analogue score | 15 minute after the block then at skin incision and "2, 6, 12, 24, and 48 hours postoperatively
  Visual analogue score at 15 minute after the block then at skin incision and "2, 6, 12, 24, and 48 hours postoperatively

SECONDARY OUTCOMES:
• Quadriceps muscle power. | In the first 48 hours after surgery.
  • Quadriceps muscle power.
Number of patients requiring analgesic rescue in the first 48 hours after surgery. | In the first 48 hours after surgery.
  Number of patients requiring analgesic rescue in the first 48 hours after surgery.
Total opioid consumption. | In the first 48 hours after surgery.
  Total opioid consumption.
Duration of the procedure | In the first 48 hours
  Duration of the procedure
Time to full anesthesia | 20 to 30 minutes before surgery
  Time to full anesthesia
Operative time | 6 hours
  Operative time
Recovery time | 48 hours after surgery
  Recovery time
Patient satisfaction questionnaire | In the first 48 hours after surgery
  Patient satisfaction
Incidence of complications | In the first 48 hours after surgery
  Incidence of complications

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University Hospital, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Li JW, Ma YS, Xiao LK. Postoperative Pain Management in Total Knee Arthroplasty. Orthop Surg. 2019 Oct;11(5):755-761. doi: 10.1111/os.12535. PMID 31663286
- [Result] Kopp SL, Borglum J, Buvanendran A, Horlocker TT, Ilfeld BM, Memtsoudis SG, Neal JM, Rawal N, Wegener JT. Anesthesia and Analgesia Practice Pathway Options for Total Knee Arthroplasty: An Evidence-Based Review by the American and European Societies of Regional Anesthesia and Pain Medicine. Reg Anesth Pain Med. 2017 Nov/Dec;42(6):683-697. doi: 10.1097/AAP.0000000000000673. PMID 29053504
- [Result] Joe HB, Choo HS, Yoon JS, Oh SE, Cho JH, Park YU. Adductor canal block versus femoral nerve block combined with sciatic nerve block as an anesthetic technique for hindfoot and ankle surgery: A prospective, randomized noninferiority trial. Medicine (Baltimore). 2016 Dec;95(52):e5758. doi: 10.1097/MD.0000000000005758. PMID 28033291
- [Result] Jensen AE, Bjorn S, Nielsen TD, Moriggl B, Hoermann R, Vaeggemose M, Bendtsen TF. Distal subsartorial compartment block of the saphenous nerve - A dissection study and a patient case series. J Clin Anesth. 2024 Feb;92:111315. doi: 10.1016/j.jclinane.2023.111315. Epub 2023 Nov 3. PMID 37926063
- [Result] Delbos A, Philippe M, Clement C, Olivier R, Coppens S. Ultrasound-guided ankle block. History revisited. Best Pract Res Clin Anaesthesiol. 2019 Mar;33(1):79-93. doi: 10.1016/j.bpa.2019.05.002. Epub 2019 May 7. PMID 31272656